CLINICAL TRIAL: NCT00796497
Title: Ondansetron Augmentation in Treatment Resistant Obsessive Compulsive Disorder: A Preliminary Single-Blind Prospective Study
Brief Title: Ondansetron in Treatment Resistant Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Neuroscience, Florence, Italy (Other)
Responsible Party: Stefano Pallanti, Institute of Neuroscience
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ONDAN-1
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; 5-ht3; ondansetron
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ondansetron (Experimental)
  Interventions: Drug: ondansetron

INTERVENTIONS:
Drug: ondansetron — ondansetron hydrochloride (oral solution) dosage of 0.25 mg twice a day for 6 weeks followed by 0,5 mg twice a day for 6 weeks for a total observation period of 12 weeks.
  Other Names: Zofran

SUMMARY:
Given that 5-HT3 receptors are indirect inhibitors of cortico-mesolimbic DA release, the 5-HT3 receptor antagonist ondansetron augmentation might potentially have efficacy in the treatment of resistant Obsessive Comulsive Disorder (OCD) patients on combined SRIs and antipsychotics.

DETAILED DESCRIPTION:
METHOD: Fourteen patients with a DSM-IV diagnosis of treatment resistant OCD, under stable treatment with SSRI's and neuroleptic augmentation will enter an 12-week single blind trial of ondansetron initiated at a dose of 0.25 mg twice daily for 6 weeks, that will be titrated to 0.5 mg twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 18 to 55
2. a Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score of ≥ 20 after ≥ 12 weeks of treatment with an established effective dose of an Selective Serotonin Reuptake Inhibitors or clomipramine and after ≥ 10 weeks of augmentation treatment with antipsychotics (risperidone at least 2 mg/day quetiapine at least 150 mg/day; olanzapine at least 5mg/day; haloperidol titrated at least 10 mg/day; aripiprazole at least 10 mg/day)

Exclusion Criteria:

1. a history of alcohol or substance abuse
2. current severe depressive symptoms, bipolar disorder, panic disorder, schizophrenia, or other psychiatric conditions
3. heart disease, arrhythmia, liver problems, including cirrhosis, seizures, glaucoma or serious medical disease
4. hoarding as only Obsessive Compulsive symptom
5. women of childbearing potential not using a medically acceptable contraceptive method.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 6th 12th week

SECONDARY OUTCOMES:
clinical global impression (CGI) | 6th e 12th

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Pallanti, MD, Principal Investigator — Istituto di Neuroscienze
Locations (1):
- Institute of Neuroscience, Florence, Italy, Italy

REFERENCES:
- [Background] Hewlett WA, Schmid SP, Salomon RM. Pilot trial of ondansetron in the treatment of 8 patients with obsessive-compulsive disorder. J Clin Psychiatry. 2003 Sep;64(9):1025-30. doi: 10.4088/jcp.v64n0907. PMID 14628977
- [Derived] Pallanti S, Bernardi S, Antonini S, Singh N, Hollander E. Ondansetron augmentation in treatment-resistant obsessive-compulsive disorder: a preliminary, single-blind, prospective study. CNS Drugs. 2009 Dec;23(12):1047-55. doi: 10.2165/11530240-000000000-00000. PMID 19958042